CLINICAL TRIAL: NCT05325034
Title: Guideline Oriented Approach To Lipid Lowering In Asia-Pacific (GOAL-ASIA)
Brief Title: Guideline Oriented Approach To Lipid Lowering In Asia-Pacific
Acronym: GOAL-ASIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stephen Nicholls (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Stephen Nicholls, Professor, Monash University
Organization: Monash University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APCMC-1
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Acute Coronary Syndrome; Atherosclerosis; Hypercholesterolemia
Keywords: Acute Coronary Syndrome; Lipid management; Cholesterol
MeSH Terms: conditions — Cardiovascular Diseases; Acute Coronary Syndrome; Atherosclerosis; Hypercholesterolemia | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Multinational, patient-level randomised, multi-phase standard-of-care control arm, parallel group, implementation study.
  Patients will be recruited during hospitalisation and be randomised to a multifaceted intervention to be delivered either 'early' (baseline) or 'late' (6 months), in a 1:1 fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early intervention (Active Comparator): Participants randomised to 'early' will receive the intervention at baseline through 6 months. while those randomised to 'late' will receive standard-of-care and represent a control arm over this period.
  Interventions: Behavioral: Early Intervention
- Late intervention (Other): Those randomised to 'late' will receive standard-of-care and represent a control arm to the early intervention group.
  Interventions: Behavioral: Early Intervention

INTERVENTIONS:
Behavioral: Early Intervention — Participant and clinician lipid score card to increase the likelihood of effecting guideline-directed change in lipid lowering therapy through two key actors - both the patient and their clinician(s).
  The Score Card documents four key fields to be completed by the participant, study team and participant's regular clinician including 1) 'current' LDL-C level, 2) participant's level of adherence to lipid-lowering therapy using modified Voil's criteria, 3) lipid-lowering management decisions made at the clinician's appointment and 4) currently prescribed lipid-lowering therapies.

SUMMARY:
Multinational, patient-level randomised, multi-phase standard-of-care control arm, parallel group, implementation study.

Patients will be recruited during hospitalisation and be randomised to a multifaceted intervention to be delivered either 'early' (baseline) or 'late' (6 months), in a 1:1 fashion.

DETAILED DESCRIPTION:
The study will be conducted over two phases.

In phase I (0-6 months), participants randomized to 'early' will receive the intervention at baseline through 6 months, while those randomized to 'late' will receive standard-of-care and represent a control arm over this period.

In phase II (6 to 12 months), those randomized to 'late' will receive the intervention at 6 months, while the 'early' group will continue in follow-up.

Multifaceted Intervention The intervention aims to increase the likelihood of effecting guideline-directed change in lipid lowering therapy through two key actors - both the patient and their clinician(s). The intervention is deliberately nested within routine clinical care to enhance the generalisability of the findings beyond a research environment and to reflect other elements of real world practice.

* Patient-and-clinician 'Cholesterol score card'. This passport-sized document will serve as a communication, engagement and activation tool for patients. It will be provided to participants at the commencement of the intervention and filled out at each study follow up visit. Participants will be encouraged to fill out sections at clinically-driven follow up appointments with their treating clinicians (e.g. general practitioner, cardiologist). The Score Card documents four key fields to be completed by the participant, study team and participant's regular clinician including 1) 'current' LDL-C level, 2) participant's level of adherence to lipid-lowering therapy using modified Voil's criteria, 3) lipid-lowering management decisions made at the clinician's appointment and 4) currently prescribed lipid-lowering therapies.
* Risk stratification for recurrent events. As part of the intervention, each participant will have their SMART Risk score of a recurrent event assessed using the 'U-prevent' online calculator. In addition, each participant's Lp(a) will be measured and presented graphically on a continuum of risk. Both of these risk assessments will be sent to the treating primary care clinician and a copy provided to the participant.

Standard of care Participants allocated to 'late' will receive standard-of-care for the first 6 months which involves the provision of the participant's lipid profile to their nominated primary care physician/general practitioner at 6 weeks, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Admission for Type I myocardial infarction

Exclusion Criteria:

* LDL <1.4mmol/L at baseline
* Unable to provide contact details of primary care physician/general practitioner
* Unable to provide written informed consent.
* Unlikely to survive >12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving an LDL <1.4mmol/L | 6 months
  Proportion of patients achieving an LDL <1.4mmol/L at 6 months. This will be determined from values obtained through local laboratory testing.

SECONDARY OUTCOMES:
Proportion of patients who undergo intensification of lipid-lowering therapy | 6 months
  Proportion of patients who undergo intensification of lipid-lowering therapy in 6 months
Proportion of patients prescribed high-intensity statin | 6 months
  Proportion of patients prescribed a guideline-recommended high-intensity statin through 6 months
Proportion of patients prescribed high-intensity statin at 6 months | 6 months
  Proportion of patients prescribed a guideline-recommended high-intensity statin at 6 months
Adherence to lipid lowering therapy | 6 months
  Proportion of patients reporting high levels of adherence to their lipid lowering therapy at 6 months
Patient activation and engagement in care | 6 months
  Level of patient activation and engagement in their care at 6 months compared with baseline
Proportion of patients achieving LDL<1.4mmol/L at 12 months | 12 months
  Proportion of patients achieving LDL<1.4mmol/L at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nicholls, MBBS, PhD, Principal Investigator — Monash University
Locations (22):
- Australia (5):
  - Illawarra Shoalhaven Local Health District, Wollongong, New South Wales
  - Cairns & Hinterland Hospital & Health Service, Cairns, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Health, Clayton, Victoria
  - Western Health, Melbourne, Victoria
- Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning, China
- All India Institute of Medical Sciences, New Delhi, India
- Japan (4):
  - Fukuoka University Hospital, Fukuoka
  - Kyorin University Hospital, Mitaka
  - National Cerebral and Cardiovascular Center, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Osaka
- Malaysia (3):
  - University Teknologi MARA, Hospital UiTM, UiTM Medical Centre, Shah Alam, Selangor
  - National Heart Institute, Kuala Lumpur
  - University of Malaysia Medical Centre, Kuala Lumpur
- Singapore (2):
  - National Heart Centre, Singapore
  - National University Hospital Singapore (NUHS), Singapore
- South Korea (2):
  - PyeongChon Hallym University Sacred Heart Hospital, Pyeongchon, Gyeonggi Province
  - Kangnam Hallym University Sacred Heart Hospital, Seoul
- National Cheng Kung University Hospital, Tainan, Taiwan
- Thailand (3):
  - Siriraj Hospital, Bangkok
  - Srinagarind Hospital and Queen Sirikit Heart Center of the Northeast, Khon Kaen
  - Songklanagarind Hospital, Songkhla

IPD SHARING:
Plan to Share IPD: No